CLINICAL TRIAL: NCT00462007
Title: Efficacy and Safety of Stalevo® in Subjects With Early Wearing-off Identified Using a Screening Tool WOQ-9; an Open, Non-randomised, Multinational, Multicentre 6-week Direct Switch Study in Levodopa-treated Parkinson's Disease Patients
Brief Title: Study to Evaluate Initiation of Stalevo in Early Wearing-off
Acronym: SENSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Liisa Luotonen, Orion Pharma
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2939117
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Stalevo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Stalevo
  Interventions: Drug: Stalevo

INTERVENTIONS:
Drug: Stalevo — Oral 3-4 daily doses for 6 weeks

SUMMARY:
An open, non-randomised, multinational, multicentre direct switch study in levodopa-treated Parkinson's disease patients suffering from early wearing-off in Parkinson's disease. The study will consist of 2 consecutive periods: screening period and study treatment period. Duration of the study will be up to 8 weeks for each subject. The study treatment dosage will be determined by the subject's current, separately administered standard levodopa/DDCI treatment (3-4 doses per day, maximum of total daily dose of 600 mg levodopa) which will be switched to an equivalent dose of Stalevo® without changing the number of doses per day. The levodopa daily dose during Stalevo® treatment may be adjusted according to the study subject's clinical response.

DETAILED DESCRIPTION:
See 'Brief summary'.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with idiopathic Parkinson's disease and early wearing-off symptoms treated with standard levodopa/DDCI treatment
* Age >35 - years
* Hoehn and Yahr stage 1-3 performed during the 'ON'-stage
* At least 1 symptom identified by WOQ-9
* Dosing frequency of 3-4 doses of standard-release levodopa/DDCI (maximum total daily dose of 600 mg of levodopa)

Exclusion Criteria:

* Atypical or symptomatic Parkinson's disease
* Unpredictable OFF-periods
* Any peak-dose dyskinesia. 'OFF'-state dystonia is allowed
* Use of any rescue medications to treat symptoms of 'OFF'-state. 1 dose of soluble levodopa/DDCI is allowed.
* Concomitant treatment with non-selective monoamine oxidase (MAO) inhibitor or simultaneous use of higher than recommended doses of MAO-A and MAO-B inhibitors (selegiline 10 mg or rasagiline 1 mg allowed) or use of apomorphine.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression of Change (Patient) | 6 weeks

SECONDARY OUTCOMES:
Clinical Global Impression of Change (Investigator); United Parkinson's Disease Rating Scale (II, III); Quality of Life Visual Analogue Scale; Wearing-off Questionnaire with 9 symptoms | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang H. Oertel, Professor, Principal Investigator — Universitätsklinikum Giessen und Marburg GmbH
Locations (20):
- Germany (14):
  - Humboldt Universität Charité Neurologische Klinik, Berlin
  - St. Josef-Hospital, Klinikum der Ruhr-Universität-Bochum Neurologische Klinik, Bochum
  - Pharmakologisches Studienzentrum Chemnitz, Chemnitz
  - Nervenarztpraxis Dr Alexander Nass, Cologne
  - Universitätsklinikum Carl Gustav Carus Klinik und Poliklinik für Neurologie, Dresden
  - Gemeinschaftspraxis für Neurologie & Psychiatrie, Erbach im Odenwald
  - Neurologische Praxis Dr Christine Schuster, Giessen
  - Universitätskrankenhaus Eppendorf, Hamburg
  - Paracelsus-Elena Klinik, Kassel
  - Alexianer-Krankenhaus, Krefeld
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Asklepios Fachklinikum Stadtroda, Stadtroda
  - Eberhard-Karls-Universität, Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
  - Neurologische Klinik der Universität Ulm, Ulm
- Sweden (3):
  - Länsjukhuset Ryhov, Geriatriska Kliniken, Jönköping
  - Nyköpings Lasarett, Ger/Rehabkliniken, Nyköping
  - Visby lasarett, Neurologmottagningen, Visby
- United Kingdom (3):
  - The Royal Bournemouth Hospital, Department of Medicines for the Elderly, Bournemouth, Dorset
  - North Tyneside General Hospital, Department of Medicine, North Shields, Tyne and Wear
  - Royal Sussex County Hospital, Neurology Department, Brighton